CLINICAL TRIAL: NCT06455046
Title: Efficacy and Safety of AK104 Combined With Pemetrexed, Carboplatin and Recombinant Human Adenovirus 5 Injection in Advanced Recurrent Cervical Cancer: a Multicenter, Single-arm, Prospective Phase II Clinical Study
Brief Title: Efficacy and Safety of AK104 Combined With Chemotherapy and Recombinant Human Adenovirus 5 Injection in Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202220202
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 Combined With Chemotherapy and Recombinant Human Adenovirus 5 Injection (Experimental): The Combined Treatment Stage consists of AK104 at a dosage of 10 mg/kg, Pemetrexed at a dosage of 500mg/m2, Cisplatin with an AUC of 4-6 mg/mL/min, and Human Adenovirus 5 Injection. This treatment is administered every 3 weeks for a total of 4 cycles. Upon enrollment, the drugs are given in the following sequence on the first day of each combined treatment cycle: local injection of Human Adenovirus 5 Injection (d1-d5), intravenous infusion of AK104 (d1), intravenous infusion of Pemetrexed (d2), and intravenous infusion of Cisplatin (d2). The Maintenance Treatment Stage involves single-drug AK104 at a dose of 10 mg/kg every 3 weeks for a duration lasting up to two years.
  Interventions: Drug: AK104; Drug: Recombinant Human Adenovirus 5 Injection

INTERVENTIONS:
Drug: AK104 — PD-1/CTLA-4 bispecific antibody
  Other Names: Cadonilimab
Drug: Recombinant Human Adenovirus 5 Injection — Recombinant Human Adenovirus 5 Injection
  Other Names: Recombinant Human Adenovirus Type 5 Injection

SUMMARY:
In order to improve the clinical effect and find a new safe and effective treatment model for advanced recurrent cervical cancer, this study explored the efficacy level safety of pemetrexed, carboplatin, recombinant human adenovirus type 5, and AK104 regimen in recurrent and refractory advanced cervical cancer. For some patients with immune-resistant cervical cancer, combination chemotherapy and oncolytic virus therapy can promote the transformation of cold tumors into hot tumors, eliminate and then reverse the suppressor factors of immune resistance, and break the dilemma of immunotherapy drug resistance, which is a new method and strategy under immunotherapy drug resistance.

DETAILED DESCRIPTION:
The Combined Treatment Stage consists of AK104 at a dosage of 10 mg/kg, Pemetrexed at a dosage of 500mg/m2, Cisplatin with an AUC of 4-6 mg/mL/min, and Human Adenovirus 5 Injection. This treatment is administered every 3 weeks for a total of 4 cycles. Upon enrollment, the drugs are given in the following sequence on the first day of each combined treatment cycle: local injection of Human Adenovirus 5 Injection (d1-d5), intravenous infusion of AK104 (d1), intravenous infusion of Pemetrexed (d2), and intravenous infusion of Cisplatin (d2). The Maintenance Treatment Stage involves single-drug AK104 at a dose of 10 mg/kg every 3 weeks for a duration lasting up to two years.

ELIGIBILITY:
Inclusion Criteria:

- 1）Enrollees in this study will be voluntary participants who sign a written informed consent form and are capable of adhering to scheduled visits and related procedures.2) Ages between 18 and 75 years old.3) Histologically or cytologically confirmed cases of persistent, recurrent, or metastatic cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma. Note: A pathological report is necessary for confirmation of the original primary tumor histology.4) Must have experienced failure with at least one standard systemic treatment and documented disease progression: Failure is defined as progression or recurrence within six months after at least one cycle of standard systemic treatment. Patients who have developed immune acquired resistance may also be included if they experienced PD after achieving CR or PR with anti-PD-1/PD-L1 antibody treatment, or PD after experiencing SD≥6 months with anti-PD-1/PD-L1 antibody treatment.

5) Not suitable for local treatments such as unresectable surgery and/or definitive concurrent radiotherapy and chemotherapy.6) The interval between the end of previous systemic treatment and the first dose of the study drug must be ≥2 weeks. Additionally, any treatment-related adverse events must have recovered to a grade ≤1 according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0 (excluding hair loss and fatigue).7) At least one measurable target lesion must be present according to RECIST V1.1 criteria.8）At least one lesion that can receive local injection therapy using recombinant human adenovirus type 5 should also meet RECIST V1.1 criteria as a measurable lesion.9) ECOG PS 0 or 1.10) The anticipated survival time should be ≥12 weeks.11) Female subjects of reproductive age are required to use effective contraception throughout the treatment period and for at least 5 months after their final dose of the investigational drug.12) Participants must consent to providing an adequate amount of tumor tissue samples for PD-L1 expression detection, which may include archived tumor samples such as paraffin blocks or a sufficient number of unstained slides meeting the study's detection requirements. If no archived tumor tissue samples are available, participants agree to undergo biopsy of the tumor lesion.13）With good organ and hematopoietic function.

Exclusion Criteria:

- 1) Diagnosed with other malignancies within the 5 years preceding initial dosing, excluding surgically cured basal cell carcinoma or squamous cell carcinoma of the skin, in situ carcinoma that has been surgically resected, and/or papillary thyroid carcinoma. Subjects with histologically confirmed small cell (neuroendocrine) cervical cancer, cervical sarcoma, and gastric-type cervical adenocarcinoma.2) Infection at the injection site.3) Presence of ascites, pleural effusion, or pericardial effusion accompanied by clinical symptoms or necessitating drainage. Subjects without clinical symptoms or requiring drainage who have ceased drainage for a minimum of 3 days and show no significant increase in fluid accumulation may be included.4) Individuals scheduled for or having undergone organ or bone marrow transplantation previously.5) Acute or chronic active hepatitis B or C infection with HBV DNA >200IU/ml or 103 copies/ml; positive anti-HCV antibody and HCV-RNA level above detection limit. Those treated with nucleoside analog antiviral agents resulting in HBV DNA/HCV-RNA levels below specified standards can be included.

6) Central nervous system (CNS) metastasis involving meningeal metastasis or symptomatic CNS metastasis. Asymptomatic brain metastases patients showing stable symptoms after treatment for at least 2 weeks may participate if they meet specific criteria: measurable lesions outside the CNS; absence of meningeal/midbrain/pons/cerebellum/medulla oblongata/spinal cord metastases; no history of intracranial hemorrhage; cessation of hormone therapy 14 days before first dose.7）Any life-threatening bleeding event within the past three months including need for blood transfusion，surgery，local treatment，or ongoing medication therapy.8）Arterial thrombosis，embolism，or ischemia within six months prior to enrollment including myocardial infarction，unstable angina pectoris ，cerebrovascular accident etc。A history of deep vein thrombosis（DVT）or any other serious thromboembolic events within three months prior to enrollment are not considered "serious" thromboembolic events.9）Hepatic vein thrombosis involving both hepatic portal trunk & left/right branches；hepatic portal trunk & mesenteric superior/inferior veins；superior vena cava thrombosis/superior vena cava syndrome.10）Tumor invasion into important surrounding organs/blood vessels such as great mediastinal vessels/superior vena cava/inferior vena cava/abdominal aorta/iliac vessels/trachea/esophagus；risk of tracheoesophageal fistula /mediastinal pleural fistula development.11）Uncontrollable hypertension defined as systolic blood pressure ≥150mmHg/diastolic blood pressure ≥100mmHg/history hypertension crisis/hypertensive encephalopathy.12）Symptomatic congestive heart failure(NYHA class II-IV)/symptomatic/poorly controlled arrhythmias/prolonged QT interval(QTcF>470ms).13）Severe bleeding tendency/coagulation dysfunction/currently receiving thrombolytic therapy.14）History gastrointestinal perforation/fistula last six months/bowel obstruction(including incomplete bowel obstruction requiring parenteral nutrition)/inflammatory bowel disease/extensive bowel resection(Crohn's disease/ulcerative colitis/chronic diarrhea).15 ) History interstitial pneumonitis/drug-induced pneumonitis/radiation pneumonitis/idopathic pneumonitis /active pneumonitis.16 ) Active tuberculosis(TB)，currently receiving anti-TB therapy/or received study drug previous year.17 ) Human immunodeficiency virus(HIV)(HIV1/HIV2 antibody positive), known active syphilis infection.18 ) Active/severely uncontrolled infections hospitalization severe infections(infections/sepsis/severe pneumonia complications etc.)within four weeks prior to first dose.19 ) Oral/intravenous therapeutic antibiotics one week before starting study treatment.20 ) Systemic autoimmune diseases/requiring systemic treatment/two-year history(white vitiligo、psoriasis、alopecia、Graves' disease not requiring systemic treatment/hypothyroidism only needing thyroid hormone replacement/type1 diabetes only needing insulin replacement). Known primary immunodeficiency history Only patients with positive autoimmune antibodies need confirmation by investigator presence autoimmune disease.21 ) Immunosuppressive drugs use four weeks except nasal inhalant local corticosteroids/systemic corticosteroids physiological doses(no more than prednisone equivalent daily doses other cortico steroids temporary use relief breathing difficulties due asthma/COPD).22 ) Live attenuated vaccine four weeks planned during study period.23 ) System immune stimulant treatments four weeks.24)Major surgery(craniotomy/thoracotomy/laparotomy)prior four weeks/unhealed wound ulcer fracture.25)Uncontrolled/metabolic disorder/non-malignant organ/systemic diseases/cancer-related complications/higher medical risk uncertainty survival period evaluation.26) Other acute chronic conditions psychiatric disorders laboratory test abnormalities increasing risk participating study/receiving study drug interfering interpretation results determined investigator patient eligible participate thisstudy.27) Received oncolytic virus therapy past received anti-CTLA-4 antibodytherapy past.28) Known allergic AK104,pemetrexed,cisplatin,and Recombinant Human Adenovirus 5 Injection components/severe allergic reaction monoclonal antibodies past.29) Received investigational drug treatment previousfourweeks starting studytreatment.30) No anticancer therapies received previousfourweeks startingstudyoral chemotherapy(two-week washout oral fluoropyrimidine-based drugs), endocrine targeted therapies(small molecule targeted therapies two-week half-life longer),immunotherapy,tumor embolization Chinese herbal medicine indications.31) Pregnant breastfeeding femalepatients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
ORR | 2years
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | 2years
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Qin Xu, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China